CLINICAL TRIAL: NCT06639568
Title: Perceptions on Telemedicine Adoption in Older Adults After Major Colorectal Surgery: A Qualitative Study
Brief Title: Telemedicine Adoption in Older Adults After Major Surgery: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Pang Ning Qi, Consultant, National University Health System, Singapore
Other Study IDs: 2020/01288
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Telemedicine
Keywords: telemedicine; older adults; cancer; post-operative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview participants

SUMMARY:
The participants are invited to participate in a research study. It is important to the investigators that the participants first take time to read through and understand the information provided in this sheet. Nevertheless, before the participants take part in this research study, the study will be explained to the participants and the participants will be given the chance to ask questions. After the participants are properly satisfied that they understand this study, and that they wish to take part in the study, they must sign this informed consent form. The participants will be given a copy of this consent form to take home with them.

Telemedicine is the use of technology for patients to communicate with doctors and healthcare professionals without visiting the hospital/clinic personally. In colorectal cancer (CRC) care, telemedicine has been suggested for post-surgery follow-up via telephone consultations and video consultation. Although telemedicine is increasingly being adopted as an alternative to long-term healthcare, little is known about the acceptability of such remote care alternatives by CRC patients in Singapore.

The participants are invited because they underwent surgery for colorectal cancer 1 to 4 years ago, are Singaporean or permanent resident of Singapore and 65 years and above. As such, the investigators want to find out about the participants' knowledge, barriers and perceptions toward the use of telemedicine as an alternative to their existing CRC care.

DETAILED DESCRIPTION:
If the participants take part in this study, they will be invited to participate in an interview. They will be asked to share about what they know about teleconsultations and what they feel/think about using telemedicine services to manage their cancer surveillance. This will allow the investigators to have an in-depth understanding of their attitudes towards telemedicine. The interview will be conducted by a trained research assistant, either in a clinical consultation room for their privacy or over the phone. The interview will be audio-recorded for data analysis and will take approximately 20-25 minutes in a single session. During the interview, the investigators will not mention the participants by name but will be using salutations to address them. The investigators will also collect the participants' basic personal information (e.g., age, gender) on a demographic form for data analysis.

We will also access your medical records for your personal medical history, as well as clinical data including your disease staging, date of diagnosis, surgery details and treatment received. The information accessed will start from your first admission to NUH for CRC till the completion of any adjuvant treatment and/or CRC-related treatment. The information will subsequently be coded and be made known only to the study team for data analysis.

Any individually-identifiable data obtained during the course of this study will be stored and analysed for the purposes of this study and will not be used for future biomedical research. The participants' participation in the study will last for a single session of approximately 20 to 25 minutes. They will only be required to participate in a single interview. They will not be required to make an additional trip back to NUH to participate in this study. The interview will be administered either during their routine follow up visits or over the phone, depending on their preference. No additional cost will need to be borne by them.

ELIGIBILITY:
Inclusion Criteria:

* Study participants aged ≥65 years who had undergone surgical resection for CRC within the past 1 - 4 years at the National University Hospital in Singapore

Exclusion Criteria:

* NA

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study participants aged ≥65 years who had undergone surgical resection for CRC within the past 1 - 4 years at the National University Hospital in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Baseline
  This is a qualitative study guided by a questionnaire, hence there is no objective primary outcome measure or scale that is used

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No